CLINICAL TRIAL: NCT02298556
Title: A Prospective Noninterventional, Observational Study to Describe the Effectiveness of Angiotensin Converting Enzyme Inhibitor and Non-dihydropyridine Calcium Channel Blocker Single Pill Combination in the Management of Hypertensive Patients With Elevated Heart Rate and Type 2 Diabetes Mellitus
Brief Title: An Observational Study to Describe the Effectiveness of Angiotensin Converting Enzyme Inhibitor and Calcium Channel Blocker Combination in the Management of Hypertensive Patients With Elevated Heart Rate and Type 2 Diabetes
Acronym: HARVEST-TR
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: MonitorCRO (Industry)
Responsible Party: Sponsor
Other Study IDs: GSS-13-0019
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Hypertension; Diabetes Mellitus; ACE Inhibitors; Calcium Channel Blockers
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive patients: Hypertensive patients with elevated heart rate and type 2 diabetes mellitus

SUMMARY:
To describe the effectiveness of angiotensin-converting enzyme inhibitor and non-dihydropyridine calcium channel blocker single pill combination on systolic blood pressure (SBP) lowering in hypertensive patients with elevated heart rate and type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥ 18 years old
* Has been already diagnosed with hypertension
* Has been already diagnosed with type 2 diabetes mellitus
* Started using angiotensin-converting enzyme inhibitor and non-dihydropyridine calcium channel blocker single pill combination within a maximum of 1 week before enrolment
* Heart rate ≥70 beat per minute

Exclusion Criteria:

* Pregnant or breast feeding female
* Current need to use any other antihypertensive drug(s) in addition to angiotensin-converting enzyme inhibitor and non-dihydropyridine calcium channel blocker single pill combination
* Having any contraindication for angiotensin-converting enzyme inhibitor or non-dihydropyridine calcium channel blocker;
* Has been treated by any anti-hypertensive treatment(s) before angiotensin-converting enzyme inhibitor and non-dihydropyridine calcium channel blocker single pill combination
* Is currently participating in another clinical or non-clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: State Hospital
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Absolute change in systolic blood pressure | from baseline to week 8
  mmHg

SECONDARY OUTCOMES:
Absolute change in diastolic blood pressure (DBP) | from baseline to week 8
  mmHg
Ratio of patients achieving blood pressure ≤ 140 and/or 90 mmHg | from baseline to week 8
Ratio of responder patients (reduction of SBP ≥20 mmHg and/or DBP ≥10 mmHg) | from baseline to week 8
Absolute change of heart rate | from baseline to week 8
  beat/min
Correlation between absolute change in blood pressure and absolute change in heart rate | from baseline to week 8
The absolute change in PR interval on electrocardiography | from baseline to week 8
  ms. The PR interval indicates "atrioventricular conduction time".
The absolute change in HbA1c (if available) | from baseline to week 8
The absolute change in microalbuminuria (if available) | from baseline to week 8
  mg/mmol
The ratio of patients experiencing an adverse event including the nature of the adverse event/severe adverse event | from baseline to week 8
The correlation between physician's office and home blood pressure measurements (Difference in medians) | from baseline to week 8
  mmHg
Blood pressure variability (daily or hourly) in home blood pressure measurement | from baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Enver Atalar, Prof. Dr., Principal Investigator — Hacettepe University Faculty of Medicine Hospital Cardiology Clinic
Locations (23):
- Turkey (Türkiye) (23):
  - Research facility ID ORG-001108, Adana
  - Research facility ID ORG-001030, Ankara
  - Yıldırım Beyazıt University Yenimahalle Training and Research Hospital, Ankara
  - Research facility ID ORG-001111, Antalya
  - Research facility ID ORG-001120, Aydin
  - Research facility ID ORG-001119, Aydin
  - Research facility ID ORG-001116, Balıkesir
  - Research facility ID ORG-001112, Burdur
  - Research facility ID ORG-001123, Çorum
  - Erzurum Regional Training and Research Hospital, Erzurum
  - Atatürk University Aziziye Research Hospital, Erzurum
  - Research facility ID ORG-001118, Istanbul
  - Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - Research facility ID ORG-001117, Istanbul
  - Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi Training and Research Hospital, Istanbul
  - Research facility ID ORG-001125, Istanbul
  - Research facility ID ORG-001113, Karabük
  - Research facility ID ORG-001110, Konya
  - Research facility ID ORG-001115, Kırıkkale
  - Research facility ID ORG-001122, Trabzon
  - Uskudar PublicHospital, Üsküdar
  - Yalova Public Hospital, Yalova
  - Research facility ID ORG-001124, Zonguldak

REFERENCES:
- [Derived] Atalar E, Eskin F, Tugtekin HB, Karabulut A, Kanyilmaz S, Kirbiyik H, Ozyildiz AG. A Prospective Noninterventional, Observational Study to Describe the Effectiveness and Safety of Trandolapril and Verapamil Single-Pill Combination in the Management of Patients with Hypertension and Type 2 Diabetes Mellitus: A Harvest TR Study. Biomed Res Int. 2020 Sep 5;2020:2123601. doi: 10.1155/2020/2123601. eCollection 2020. PMID 32964020